CLINICAL TRIAL: NCT02345096
Title: A Randomized, Double-blind, Placebo Controlled Study to Evaluate the Effect of Saccharomyces Cerevisiae on Improving the Effectiveness of Conventional Treatment of Vulvo-vaginal Candidiasis
Brief Title: Effect of Saccharomyces Cerevisiae on Improving the Effectiveness of Conventional Treatment of Vulvo-vaginal Candidiasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Lesaffre International (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OP090414.LES
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Vulvo-vaginal Candidiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saccharomyces cerevisiae CNCM I-3856 (Active Comparator): In this arm, subjects will be asked to consume one capsule of Saccharomyces cerevisiae CNCM I-3856 per day.
  Interventions: Dietary Supplement: Saccharomyces cerevisiae
- placebo (Placebo Comparator): In this arm, subjects will be asked to consume one capsule of placebo per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Saccharomyces cerevisiae
  Arms: Saccharomyces cerevisiae CNCM I-3856
Dietary Supplement: Placebo
  Arms: placebo

SUMMARY:
This study aims to evaluate the effect of a specific strain of Saccharomyces cerevisiae on improving the effectiveness of conventional treatment of vulvo-vaginal candidiasis. This is a randomized, double-blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female patient with a clinical diagnosed vulvo-vaginal candidiasis
* Regularly menstruating women with normal gynaecological status
* Patient must use a contraception method
* Having given a written informed consent prior to selection
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Tumors in the genital tract or beast.
* Hypersensitivity to the study product.
* Uterine or vaginal bleeding of unknown origin.
* Use of systemic or intravaginal antibiotic or antifungal agents in the previous 14 days.
* Concomitant medication with antimycotics for other diagnoses.
* Woman with known transmitted infections such as Neisseria gonorrhoea, Chlamydia trachomatis, Treponema pallidum, herpes simplex, Trichomonas vaginalis, human papilloma virus, HIV 1 or 2.
* Immunocompromised individuals.
* Subjects not willing to stop taking probiotics in the form of dietary supplements or convenient goods
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development.
* Subject under administrative or legal supervision.
* Subject who participate to a previous study within 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Enumeration of Candida albicans in a vaginal sampling | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cherbut, MD, Principal Investigator — Independant gynecologist
Locations (1):
- Eurofins Optimed, Gières, France